CLINICAL TRIAL: NCT02692469
Title: Laparoscopic Single-Anastomosis Duodenal-Jejunal Bypass With Sleeve Gastrectomy vs Laparoscopic Duodenal Switch as a Primary Bariatric Procedure. 5 Year Patient Follow
Brief Title: Laparoscopic Single-Anastomosis Duodenal-Jejunal Bypass With Sleeve Gastrectomy vs Laparoscopic Duodenal Switch
Acronym: DSvsSADI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Dennis Hong MD, Principal Investigator, General Surgeon, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1366
Record Dates: First submitted 2016-02-03; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: Bariatric Surgery, Obesity, Laparoscopy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duodenal Switch Surgical Intervention (Active Comparator): a DS procedure involves creating a sleeve gastrectomy with preservation of the pylorus, and creation of a Roux limb with a short common channel
  Interventions: Procedure: Duodenal Switch
- Single Anastomosis Duodenal-Ileal Bypass (Experimental): The SADI defers from the DS in that after the duodenum is separated from the stomach, preserving the pylorus, a loop of bowel 200 cm from the ileo-cecal valve is anastomosed with the pylorus, thus requiring only one anastomosis
  Interventions: Procedure: Duodenal-ileal Bypass with Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Duodenal Switch — Bariatric procedure
  Other Names: DS
  Arms: Duodenal Switch Surgical Intervention
Procedure: Duodenal-ileal Bypass with Sleeve Gastrectomy — Bariatric procedure
  Other Names: SADI
  Arms: Single Anastomosis Duodenal-Ileal Bypass

SUMMARY:
Will a laparoscopic Single-Anastomosis Duodenal-ileal Bypass with Sleeve Gastrectomy produce similar or superior results when compared to a laparoscopic Duodenal Switch, as a primary surgical procedure for weight loss in bariatric patients over a 5 year period?

DETAILED DESCRIPTION:
The aims of this study are: (a) to compare SADI vs DS as a primary bariatric procedure for weight loss; (b) to compare the minor and major complications of SADI vs DS (c) to compare SADI vs DS for remission rates of type 2 diabetes (d) to compare SADI vs DS for remission rates of hypertension (e) to compare SADI vs DS for weight regain at 5 years (f) to compare SADI vs DS for metabolic alterations. The investigators hypothesize that both procedures will have similar weight loss and metabolic remission results. If the complication rates of SADI are similar or superior to the complication rates of the DS, then the investigators could propose the SADI as a viable alternative to the DS in patients with high BMIs requiring increased weight loss.

The investigators will conduct a prospective randomized study. The study will include 140 patients who are scheduled for bariatric procedures. The patients will be stratified into 2 groups. The first group will continue according to the standard bariatric preoperative protocol and will be assigned to a DS. The second group will also follow standard bariatric preoperative protocol but will be assigned to a SADI. Follow up of all patients will continue according to the usual bariatric clinic guidelines.

From literature, the mean excess body weight loss is 77.65% with standard deviation of 21% for Duodenal Switch bariatric surgery. If there is in truth no difference between the Duodenal Switch and SADI for excess body weight loss, then 140 patients (70 per group) are required to have 80% power for the lower limit of a one-sided 97.5% confidence interval (or equivalently a 95% two-sided confidence interval) will be above the non-inferiority limit of -10%.

Participants must meet ALL of the following inclusion criteria:

* Fulfilled criteria for bariatric surgery as coined by National Institutes of Health.
* Their age is ≥18 years and ≤70 years
* Able and willing to give written consent

Participants who meet any of the following criteria at the time of the baseline visit are NOT eligible to be enrolled in this study:

* Contra-indication to general anesthesia
* Any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Pregnant or lactating female (Women of child bearing potential must take a pregnancy test prior to surgery)
* History of alcohol abuse (>30 g/day in men or >20 g/day in women)

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet ALL of the following inclusion criteria:

  * Fulfilled criteria for bariatric surgery as coined by National Institutes of Health.
  * Their age is ≥18 years and ≤70 years
  * Able and willing to give written consent

Exclusion Criteria:

* Participants who meet any of the following criteria at the time of the baseline visit are NOT eligible to be enrolled in this study:

  * Contra-indication to general anesthesia
  * Any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
  * Pregnant or lactating female (Women of child bearing potential must take a pregnancy test prior to surgery)
  * History of alcohol abuse (>30 g/day in men or >20 g/day in women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Excess weight loss | 5 years
  BMI and body weight will be measured and compared to preoperative reference values

SECONDARY OUTCOMES:
Remission of type 2 diabetes | 5 years
  The presence and remission of type 2 diabetes will be diagnosed according to the American Diabetes Association's current criteria:
  1. A1C ≥6.5 percent, OR
  2. FPG ≥126 mg/dL (7.0 mmol/L), OR
  3. Two-hour plasma glucose ≥200 mg/dL (11.1 mmol/L) during an OGTT, OR
  4. In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dL (11.1 mmol/L).
Remission of hypertension | 5 years
  The presence and remission of hypertension will be diagnosed by the definitions suggested in 2003 by the seventh report of the Joint National Committee (JNC 7) and are based upon the average of two or more properly measured readings at each of two or more office visits after an initial screen:
  * Normal blood pressure: systolic <120 mmHg and diastolic <80 mmHg
  * Prehypertension: systolic 120 to 139 mmHg or diastolic 80 to 89 mmHg (see "Prehypertension")
  * Hypertension:
    * Stage 1: systolic 140 to 159 mmHg or diastolic 90 to 99 mmHg
    * Stage 2: systolic ≥160 mmHg or diastolic ≥100 mmHg
Surgical complications | 1 year
  According to the Clavien-Dindo Classification of surgical complications
Metabolic alterations | 5 years
  Blood levels will be measured pre-operatively a on a regular schedule after surgery for:
  zinc, magnesium, phosphate, albumin, PTH, HbA1C, ferritin, calcium, Iron binding capacity, total proteins, Hb, Cholesterol levels, LDL, Vit. D, Vit. A and Vit. B12 to ensure they are in normal range.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hong, MD FRCSC, Principal Investigator — St. Joseph Healthcare Hamilton, McMaster University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sanchez-Pernaute A, Rubio Herrera MA, Perez-Aguirre E, Garcia Perez JC, Cabrerizo L, Diez Valladares L, Fernandez C, Talavera P, Torres A. Proximal duodenal-ileal end-to-side bypass with sleeve gastrectomy: proposed technique. Obes Surg. 2007 Dec;17(12):1614-8. doi: 10.1007/s11695-007-9287-8. Epub 2007 Nov 27. PMID 18040751
- [Result] Sanchez-Pernaute A, Herrera MA, Perez-Aguirre ME, Talavera P, Cabrerizo L, Matia P, Diez-Valladares L, Barabash A, Martin-Antona E, Garcia-Botella A, Garcia-Almenta EM, Torres A. Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S). One to three-year follow-up. Obes Surg. 2010 Dec;20(12):1720-6. doi: 10.1007/s11695-010-0247-3. PMID 20798995
- [Result] Sanchez-Pernaute A, Rubio MA, Perez Aguirre E, Barabash A, Cabrerizo L, Torres A. Single-anastomosis duodenoileal bypass with sleeve gastrectomy: metabolic improvement and weight loss in first 100 patients. Surg Obes Relat Dis. 2013 Sep-Oct;9(5):731-5. doi: 10.1016/j.soard.2012.07.018. Epub 2012 Aug 7. PMID 22963820
- [Result] Sovik TT, Taha O, Aasheim ET, Engstrom M, Kristinsson J, Bjorkman S, Schou CF, Lonroth H, Mala T, Olbers T. Randomized clinical trial of laparoscopic gastric bypass versus laparoscopic duodenal switch for superobesity. Br J Surg. 2010 Feb;97(2):160-6. doi: 10.1002/bjs.6802. PMID 20035530